CLINICAL TRIAL: NCT07097142
Title: The Phase III Adaptive Radiation and Chemotherapy for Muscle Invasive Bladder Cancer Trial (ARCHER)
Brief Title: Testing Shorter Duration Radiation Therapy Versus the Usual Radiation Therapy in Patients Receiving the Usual Chemotherapy Treatment for Bladder Cancer, ARCHER Study
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-GU015; NCI-2025-04136 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GU015 (Other: NRG Oncology); NRG-GU015 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2025-07-21; First posted 2025-07-31 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Muscle Invasive Bladder Urothelial Carcinoma; Stage II Bladder Cancer AJCC v8; Stage IIIA Bladder Cancer AJCC v8
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Specimen Handling; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Fluorouracil; dehydroftorafur; Gemcitabine; Radiation Dose Hypofractionation; Radiation; Magnetic Resonance Spectroscopy; Mitomycin; Mitozytrex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (hypofractionated radiation therapy) (Active Comparator): Patients receive hypofractionated RT QD, Monday to Friday, for 20 treatments in the absence of disease progression or unacceptable toxicity. Patients also receive one of 3 systemic chemotherapy regimens per treating physician's choice: 1) cisplatin IV weekly for 4 weeks; 2) gemcitabine IV on days 1, 4, 8, 11, 15, 18, 22 and 25 or weekly for 4 weeks; or 3) mitomycin-C IV on day 1 and 5 FU, over 120 hours on days 1-5 and 22-26. Treatment is given in the absence of disease progression or unacceptable toxicity. Patients also undergo CT scan and/or MRI or FDG PET throughout the study. In addition, patients may undergo optional blood and urine sample collection throughout the study, as well as an optional biopsy during cystoscopy during follow up.
  Interventions: Procedure: Biospecimen Collection; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Fluorouracil; Drug: Gemcitabine; Radiation: Hypofractionated Radiation Therapy; Procedure: Magnetic Resonance Imaging; Drug: Mitomycin; Procedure: Positron Emission Tomography; Other: Survey Administration
- Arm II (Ultrahypofractionated radiation therapy) (Experimental): Patients receive ultra-hypofractionated RT QD, no more than twice weekly, for 5 treatments in the absence of disease progression or unacceptable toxicity. Patients also receive one of 3 systemic chemotherapy regimens per treating physician's choice: 1) cisplatin IV weekly for 4 weeks; 2) gemcitabine IV on days 1, 4, 8, 11, 15, 18, 22 and 25 or weekly for 4 weeks; or 3) mitomycin-C IV on day 1 and 5 FU, over 120 hours on days 1-5 and 22-26. Treatment given in the absence of disease progression or unacceptable toxicity. Patients also undergo CT scan and/or MRI or FDG PET throughout the study. In addition, patients may undergo optional blood and urine sample collection throughout the study, as well as an optional biopsy during cystoscopy during follow up.
  Interventions: Procedure: Biospecimen Collection; Drug: Cisplatin; Procedure: Computed Tomography; Drug: Fluorouracil; Drug: Gemcitabine; Procedure: Magnetic Resonance Imaging; Drug: Mitomycin; Procedure: Positron Emission Tomography; Other: Survey Administration; Radiation: Ultrahypofractionated Radiation Therapy

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood, tissue, and urine sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd; Difluorodeoxycytidine
Radiation: Hypofractionated Radiation Therapy — Undergo hypofractionated radiation therapy
  Other Names: Hypofractionated; Hypofractionated Radiotherapy; hypofractionation; Radiation, Hypofractionated
  Arms: Arm I (hypofractionated radiation therapy)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Mitomycin — Given IV
  Other Names: Ametycine; Jelmyto; MITO; Mito-C; Mito-Medac; Mitocin; Mitocin-C; Mitolem; Mitomycin C; Mitomycin pyelocalyceal; Mitomycin-C; Mitomycin-X; Mitomycine C; Mitosol; Mitozytrex; Mutamycin; Mutamycine; NCI-C04706
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Survey Administration — Ancillary studies
Radiation: Ultrahypofractionated Radiation Therapy — Undergo ultrahypofractionated radiation therapy.
  Other Names: Ultrahypofractionated Radiotherapy
  Arms: Arm II (Ultrahypofractionated radiation therapy)

SUMMARY:
This phase III trial compares the effect of decreased number of radiation (ultra-hypofractionated) treatments to the usual radiation number of treatments (hypofractionation) with standard of care chemotherapy, with cisplatin, gemcitabine or mitomycin and 5-fluorouracil for the treatment of patients with muscle invasive bladder cancer. Hypofractionated radiation therapy delivers higher doses of radiation therapy over a short period of time. Ultra-hypofractionated radiation therapy delivers radiation over an even shorter period of time than hypofractionated radiation therapy. Cisplatin is in a class of medications known as platinum-containing compounds. It works by killing, stopping or slowing the growth of tumor cells. Gemcitabine is a chemotherapy drug that blocks the cells from making DNA and may kill tumor cells. Chemotherapy drugs, such as mitomycin-C and 5-fluorouracil (5-FU), work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving ultra-hypofractionated radiation may be equally effective as hypofractionated therapy for patients with muscle invasive bladder cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Demonstrate non-inferiority of ultra-hypofractionated (stereotactic body radiation therapy [SBRT]) compared to hypofractionated radiation therapy (RT) with a 10% non-inferiority margin (from 50% to 40%) in the rate of bladder-intact event-free survival (BI-EFS) at 3 years (corresponding to a hazard ratio < 1.32).

SECONDARY OBJECTIVES:

I. Compare the rates of urinary and bowel toxicity, patient-reported outcomes (PRO), event-free survival (EFS), metastasis-free survival (MFS), and overall survival (OS) between the two treatment arms.

II. Compare and evaluate symptomatic adverse events and quality of life measures that are most meaningful to patients.

III. Evaluate circulating tumor deoxyribonucleic acid (ctDNA) as a biomarker to determine whether it is predictive of disease recurrence and as a secondary outcome variable.

EXPLORATORY OBJECTIVES:

I. Evaluate ctDNA, tissue-free minimal residual disease (tfMRD) and urine tumor DNA (utDNA) as biomarkers for predicting recurrence.

II. Evaluate tfMRD, obtained at the time of progression, to determine if it captures the presence of disease.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive hypofractionated radiation therapy (RT) once daily (QD), Monday to Friday, for 20 treatments in the absence of disease progression or unacceptable toxicity. Patients also receive one of 3 systemic chemotherapy regimens per treating physician's choice: 1) cisplatin intravenously (IV) weekly for 4 weeks; 2) gemcitabine IV on days 1, 4, 8, 11, 15, 18, 22 and 25 or weekly for 4 weeks; or 3) mitomycin-C IV on day 1 and fluorouracil (5 FU), over 120 hours on days 1-5 and 22-26. Treatment is given in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) scan and/or magnetic resonance imaging (MRI) or fluorodeoxyglucose (FDG) positron emission tomography (PET) throughout the study. In addition, patients may undergo optional blood and urine sample collection throughout the study, as well as an optional biopsy during cystoscopy during follow up.

ARM II: Patients receive ultra-hypofractionated RT QD, no more than twice weekly, for 5 treatments in the absence of disease progression or unacceptable toxicity. Patients also receive one of 3 systemic chemotherapy regimens per treating physician's choice: 1) cisplatin IV weekly for 4 weeks; 2) gemcitabine IV on days 1, 4, 8, 11, 15, 18, 22 and 25 or weekly for 4 weeks; or 3) mitomycin-C IV on day 1 and 5 FU, over 120 hours on days 1-5 and 22-26. Treatment given in the absence of disease progression or unacceptable toxicity. Patients also undergo CT scan and/or MRI or FDG PET throughout the study. In addition, patients may undergo optional blood and urine sample collection throughout the study, as well as an optional biopsy during cystoscopy during follow up.

After completion of study treatment, patients are followed up at week 16, every 3 months for 3 years then every 6 months to year 5.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven, cT2-T3,N0M0 urothelial carcinoma of the bladder prior to randomization.

  * Note: Patients with mixed urothelial carcinoma will be eligible for the trial, but the presence of small cell carcinoma will make a patient ineligible
* Must undergo a transurethral resection of bladder tumor (TURBT) prior to randomization. Patients may have either completely or partially resected tumors as long as the treating urologist attempted maximal resection
* Must undergo radiological staging prior to randomization. Imaging of chest, abdomen, and pelvis must be performed using CT or MRI (with or without contrast is acceptable). Patients must not have evidence of T4 or node positive disease. Fluorodeoxyglucose (FDG) PET imaging is acceptable for radiological staging
* If any lymph nodes ≥ 1.0 cm in shortest cross-sectional diameter are noted on imaging (CT / MRI of abdomen and pelvis), then the patient must have had a biopsy of the enlarged lymph node showing no tumor involvement prior to randomization
* No diffuse carcinoma in situ (CIS) based on cystoscopy and biopsy
* No definitive clinical or radiologic evidence of metastatic disease
* Must not have had urothelial carcinoma or histological variant at any site outside of the urinary bladder within 24 months prior to registration except Ta/T1/Carcinoma in situ (CIS) of the upper urinary tract including renal pelvis and ureter if the patient had undergone complete nephroureterectomy
* Age ≥ 18
* Zubrod performance status of ≤ 2
* Not pregnant and not nursing

  * Negative urine or serum pregnancy test (in persons of childbearing potential) within 14 days prior to registration. Childbearing potential is defined as any person who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal
* Absolute neutrophil count (ANC) ≥ 1,500 cells/mm^3
* Platelets ≥ 100,000 cells/mm^3
* Hemoglobin ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve hemoglobin [Hgb]) ≥ 8.0 g/dl is acceptable)
* Creatinine clearance (CrCL) of ≥ 30 mL/min by the Cockcroft-Gault formula
* Total bilirubin ≤ 2 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 3 x institutional ULN
* All adverse events associated with any prior therapy must have resolved to Common Terminology Criteria for Adverse Events (CTCAE) grade ≤ 3 prior to randomization
* For patients who have completed neoadjuvant therapy, they are eligible if the pre-neoadjuvant therapy diagnosis (TURBT path) is within 180 days before randomization
* Must not have had prior pelvic radiation
* New York Heart Association Functional Classification II or better (NYHA Functional Classification III/IV are not eligible) (Note: Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification.)
* No active infection requiring IV antibiotics
* Patients with hydronephrosis are eligible if they have unilateral hydronephrosis and kidney function meet criteria specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Estimated)
Dates: Start 2026-05-11 (Estimated); Primary Completion 2030-05-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Bladder-intact event-free survival (BI-EFS) | Up to 3 years
  Defined as histologically proven presence of muscle invasive bladder cancer (MIBC), radiographic evidence of nodal or metastatic disease, performance of radical cystectomy, or death from any cause. Time to event will be calculated from the date of randomization. BI-EFS will be estimated in the two treatment groups using the Kaplan-Meier method and the hazard ratio between ultra-hypofractionation and hypofractionation estimated by fitting a Cox proportional hazards regression model, including a treatment arm indicator variable and adjusting for the three stratification factors employed in the randomization.

SECONDARY OUTCOMES:
Incidence of urinary adverse events | Up to year 2
  Will be graded per Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v 5.0). The proportion of patients experiencing grade 3 or higher urinary/bowel toxicity within two years of initiation of treatment will be compared between the two treatment groups using a chi-square test. The 95% confidence interval (CI) width for the true difference will be at most ± 8.9%.
Incidence of bowel adverse events | Up to year 2
  Will be graded per CTCAE v 5.0. The proportion of patients experiencing grade 3 or higher urinary/bowel toxicity within two years of initiation of treatment will be compared between the two treatment groups using a chi-square test. The 95% CI width for the true difference will be at most ± 8.9%.
Quality of life | At baseline, 4 weeks, 16 weeks, 13 months, 25 months, and 37 months
  As measured by the Functional Assessment of Cancer Therapy-Bladder instrument.
Event free survival | From randomization to histologically proven presence of MIBC, radiographic evidence of nodal or metastatic disease, or death from any cause, up to 5 years
  Kaplan-Meier curves will be generated and the groups compared using a stratified logrank test (stratified by the randomization stratification factors). In addition, a Cox regression model will be fit, including treatment arm and the stratification factors.
Metastasis-free survival | From randomization to radiographic evidence of metastatic disease or death due to any cause, up to 5 years
  Kaplan-Meier curves will be generated and the groups compared using a stratified logrank test. A Cox regression model will also be fit, including treatment arm and the stratification factors.
Overall survival | From randomization to death from any cause, up to 5 years
  Kaplan-Meier curves will be generated and the groups compared using a stratified logrank test. A Cox regression model will also be fit, including treatment arm and the stratification factors.
Incidence of adverse events (AE) | Up to year 2
  Will be graded using CTCAE v 5.0. AE rates between the two treatment groups will be compared using chi-square or Fisher exact tests.

OTHER OUTCOMES:
ctDNA | At baseline, 4, 16, 28, 40, and 56 weeks from start of chemotherapy
  Will be analyzed as prognostic markers by fitting Cox regression models for BI-EFS.
Primary outcome treatment effect by sex | Up to 5 years
  The corresponding 95% CIs will be provided.
Primary outcome treatment effect by ethnicity | Up to 5 years
  The corresponding 95% CIs will be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Scott E Delacroix, Principal Investigator — NRG Oncology
Locations (191):
- United States (191):
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Beebe Medical Center, Lewes, Delaware
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - UM Sylvester Comprehensive Cancer Center at Doral, Doral, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - OSF Saint Anthony's Health Center, Alton, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Rush MD Anderson Cancer Center at Rush Oak Park, Oak Park, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - The Iowa Clinic PC, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Metairie, Metairie, Louisiana
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Bronson Battle Creek, Battle Creek, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo, Kalamazoo, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Henry Ford Wyandotte Hospital, Wyandotte, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - University of Kansas Cancer Center - Briarcliff, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Lake Regional Hospital, Osage Beach, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Hi-Line Sletten Cancer Center, Havre, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - UH Seidman Cancer Center at UH Avon Health Center, Avon, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - MD Anderson in The Woodlands, Conroe, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Bon Secours Cancer Institute at Reynolds Crossing, Richmond, Virginia
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin